CLINICAL TRIAL: NCT03423459
Title: CoreValve Evolut Pro Prospective Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: EPROMPT
Record Dates: First submitted 2018-01-18; First posted 2018-02-06 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- CT Cohort: 1. Compare the rate of ≥mild PVL in patients with none/mild versus moderate/severe LVOT calcification.
  2. Comparison of the rate of PPM implantation in patients with none/mild versus moderate/severe LVOT calcification.
  3. Determine how the Evolut PRO conforms to LVOT calcification.
  4. Compare the impact of LVOT calcification on the implantation depth of the Evolut PRO.
  5. Analyze the interaction and geometry of the Evolut PRO in patients with moderate/severe LVOT calcification.
  6. Assess for leaflet thickening, subclinical leaflet thrombosis and/or restricted leaflet motion 30-60 days after TAVR.
  Interventions: Device: TAVR
- Non-CT Cohort: 1. Compare the rate of ≥mild PVL with the Evolut PRO with a propensity score matched cohort of historical control subjects who underwent TAVR with the Evolut R and/or CoreValve within the MedStar Health System.
  2. Determine which features of LVOT calcification (volume, location relative to aortic annulus and sinuses, prominence into the LVOT lumen) predict ≥mild PVL.
  3. Determine which features of LVOT calcification (volume, location relative to aortic annulus and sinuses, prominence into the LVOT lumen) predict PPM implantation.
  Interventions: Device: TAVR

INTERVENTIONS:
Device: TAVR — Transcatheter Aortic Valve Replacement

SUMMARY:
The primary objective of this study is to evaluate the real-world performance of the CoreValve Evolut PRO transcatheter aortic valve, including leaflet function, in a prospective observational registry.

DETAILED DESCRIPTION:
The CoreValve Evolut PRO transcatheter aortic valve was approved by the FDA in March 2017 to treat patients with symptomatic severe aortic stenosis at high or extreme risk for open heart surgery, and in July 2017 for intermediate risk patients. This latest generation device features an outer wrap to improve annular sealing and reduce paravalvular leak.

In this observational study, baseline demographic and imaging characteristics, procedural details and clinical outcomes of patients undergoing transcatheter aortic valve replacement with the CoreValve Evolut PRO will be prospectively collected into a registry database. The institutional Heart Team will select patients according to standard practice.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic severe aortic stenosis
2. Intermediate, high or extreme surgical risk
3. The institutional Heart Team determines that transcatheter aortic valve replacement with an Evolut Pro device is appropriate

Exclusion Criteria:

1. Subject unable or unwilling to give informed consent
2. For subjects in the CT arm only, renal function precluding the administration of iodinated contrast for cardiac CT (eGFR < 30 ml/min/1.73m2). An exception to this exclusion criterion is made if the subject is established on renal replacement therapy and is therefore able to receive intravenous iodinated contrast media.
3. Pregnancy or intent to become pregnant prior to completion of all protocol follow-up procedures

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study is a prospective registry of subjects with symptomatic severe aortic stenosis undergoing TAVR with a commercially-approved self-expanding transcatheter heart valve. A subgroup of subjects will undergo additional research contrast-enhanced 4D CT at 30-60 days after TAVR. Otherwise, all additional test and TAVR implantation procedures are as per standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Device success: | 30 days
  Absence of procedural mortality Intended performance of the prosthetic heart valve (no prosthesis-patient mismatch and mean aortic valve gradient<20 mm Hg or peak velocity<3 m/s, AND no moderate or severe prosthetic valve regurgitation)
All Cause Mortality | 30 days
  all causes of death
All Stroke (disabling and non-disabling | 30 days
  Stroke will evaluated using the VARC-2 definition
Life Threatening Bleeding | 30 Days
  Life Threatening Bleeding will be evaluated using the VARC-2 definition
Acute Kidney Injury Stage 2 or 3 | 30 days
  AKI will be evaluated using the VARC-2 definition of Stage 2 or 3 AKI
Coronary Artery Obstruction requiring intervention | 30 days
  This will be assessed if by noting whether the patient has a re intervention
Major Vascular Complication | 30 days
  Major Vascular Complication will be evaluated using the VARC-2 definition of Major Vascular Complication
Valve - related Dysfunction | 30 Days
  Valve related dysfunction will be evaluated by determining whether the subject has a repeat procedure such as a BAV, TAVI, or SAVR

SECONDARY OUTCOMES:
Prosthetic valve dysfunction #1 | 1 year
  Mean aortic valve gradient ≥20 mm Hg
Prosthetic valve dysfunction #2 | 1 year
  Moderate-severe transvalvular aortic regurgitation as determined by the echo core lab
Prosthetic valve dysfunction #3 | 1 year
  Abnormal leaflet thickening on CT as determined by the CT Core lab
Prosthetic valve dysfunction #4 | 1 year
  Decreased leaflet mobility on CT as determined by the CT Core lab
Prosthetic valve dysfunction | 1 year
  Leaflet thrombosis on CT as determined by the CT Core lab
Reduction in PVL | Discharge thru to 1 year
  This will be evaluated by echo core lab findings

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Medstar Union Memorial Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merdler I, Case BC, Bhogal S, Reddy PK, Zhang C, Ali S, Gallino PE, Jackman C, Ben-Dor I, Satler LF, Cohen JE, Rogers T, Waksman R. Temporal trends with the Evolut family of self-expanding transcatheter heart valves: A single-center experience. Catheter Cardiovasc Interv. 2024 Jul;104(1):125-133. doi: 10.1002/ccd.31088. Epub 2024 May 20. PMID 38769727
- [Derived] Medranda GA, Soria Jimenez CE, Torguson R, Case BC, Forrestal BJ, Ali SW, Shea C, Zhang C, Wang JC, Gordon P, Ehsan A, Wilson SR, Levitt R, Parikh P, Bilfinger T, Hanna N, Buchbinder M, Asch FM, Weissman G, Shults CC, Garcia-Garcia HM, Ben-Dor I, Satler LF, Waksman R, Rogers T. Lifetime management of patients with symptomatic severe aortic stenosis: a computed tomography simulation study. EuroIntervention. 2022 Aug 5;18(5):e407-e416. doi: 10.4244/EIJ-D-21-01091. PMID 35321859
- [Derived] Forrestal BJ, Case BC, Yerasi C, Shea C, Torguson R, Zhang C, Ben-Dor I, Deksissa T, Ali S, Satler LF, Shults C, Weissman G, Wang JC, Khan JM, Waksman R, Rogers T. Risk of Coronary Obstruction and Feasibility of Coronary Access After Repeat Transcatheter Aortic Valve Replacement With the Self-Expanding Evolut Valve: A Computed Tomography Simulation Study. Circ Cardiovasc Interv. 2020 Dec;13(12):e009496. doi: 10.1161/CIRCINTERVENTIONS.120.009496. Epub 2020 Dec 4. PMID 33272031